CLINICAL TRIAL: NCT02055196
Title: A Phase I Study of Intracranially Administered Carboxylesterase-Expressing Neural Stem Cells in Combination With Intravenous Irinotecan in Patients With Recurrent High-Grade Gliomas
Brief Title: Genetically Modified Stem Cells and Irinotecan Hydrochloride in Treating Patients With Recurrent High-Grade Gliomas
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: New study written
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13455; NCI-2014-00117 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 13455 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2014-01-30; First posted 2014-02-05 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2014-05

CONDITIONS: Adult Anaplastic Astrocytoma; Adult Anaplastic Oligodendroglioma; Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma; Recurrent Adult Brain Tumor
MeSH Terms: conditions — Astrocytoma; Oligodendroglioma; Glioblastoma; Gliosarcoma; Brain Neoplasms | interventions — Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (neuronal stem cells, irinotecan hydrochloride) (Experimental): Patients receive carboxylesterase-expressing allogeneic neural stem cells via intracerebral catheter on day 1 of week 1; weeks 1 and 3, weeks 1, 2, and 3; or weeks 1, 2, 3, and 4. Patients also receive irinotecan hydrochloride IV over 90 minutes on day 3 of week 1; weeks 1 and 3, weeks 1, 2, and 3; or weeks 1, 2, 3, and 4. Courses repeat every 6 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: carboxylesterase-expressing allogeneic neural stem cells; Drug: irinotecan hydrochloride; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: carboxylesterase-expressing allogeneic neural stem cells — Given via intracerebral catheter
  Other Names: hCE1m6-NSC
Drug: irinotecan hydrochloride — Given IV
  Other Names: Campto; Camptosar; CPT-11; irinotecan; U-101440E
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of genetically modified stem cells when given together with irinotecan hydrochloride in treating patients with recurrent high-grade gliomas. Irinotecan hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Placing a gene that has been created in the laboratory into neural stem cells and injecting it into the brain may help irinotecan hydrochloride kill more tumor cells once it reaches the brain.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To define the recommend phase II doses of intracranially administered active modified human form of carboxylesterase (hCE1m6)- neuronal stem cells (NSCs) (carboxylesterase-expressing allogeneic neural stem cells) in combination with intravenous irinotecan (irinotecan hydrochloride).

II. To determine the biologic activity of the hCE1m6-NSCs by comparing SN-38 concentrations in the brain after treatment with hCE1m6-NSCs and irinotecan compared to irinotecan alone.

SECONDARY OBJECTIVES:

I. To investigate the relationship between hCE1m6-NSC dose and SN-38 concentrations in brain interstitium.

II. To characterize the relationship between intracerebral and systemic concentrations of irinotecan and SN-38.

III. To assess for possible development of NSC immunogenicity after first exposure and with repeat doses of NSCs.

IV. To evaluate the intracerebral distribution of NSCs by using iron-labeling as a cellular tracker.

V. To describe the clinical benefit (defined as stable disease, partial response, or complete response) in patients who receive treatment with repeat cycles of NSCs and irinotecan.

VI. To determine, at time of autopsy, the fate of the NSCs.

OUTLINE: This is a dose-escalation study of carboxylesterase-expressing allogeneic neural stem cells.

Patients receive carboxylesterase-expressing allogeneic neural stem cells via intracerebral catheter on day 1 of week 1; weeks 1 and 3, weeks 1, 2, and 3; or weeks 1, 2, 3, and 4. Patients also receive irinotecan hydrochloride intravenously (IV) over 90 minutes on day 3 of week 1; weeks 1 and 3, weeks 1, 2, and 3; or weeks 1, 2, 3, and 4. Courses repeat every 6 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for at least 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a prior, histologically-confirmed, diagnosis of a grade III or IV glioma (including glioblastoma, anaplastic astrocytoma, gliosarcoma, anaplastic oligodendroglioma, or anaplastic oligoastrocytoma), or has a prior, histologically-confirmed, diagnosis of a grade II glioma and now has radiographic findings consistent with a high-grade glioma (grade III or IV)
* Imaging studies show evidence of recurrent, supratentorial tumor(s)
* Patient's high-grade glioma has recurred or progressed after prior treatment with brain radiation and temozolomide
* Patient has a Karnofsky performance status of >= 70%
* Patient has a life expectancy of >= 3 months
* Female patients of childbearing potential and sexually-active male patients must agree to use an effective method of contraception while participating in this study; women of childbearing potential must have a negative pregnancy test =< 2 weeks prior to registration
* PROTOCOL-SPECIFIC CRITERIA
* Patient must be in need of a craniotomy for tumor resection or a stereotactic brain biopsy for the purpose of diagnosis or differentiating between tumor progression versus treatment-induced effects following radiation therapy ± chemotherapy
* Patients who will undergo tumor resection must have residual enhancing tumor (i.e. a gross total resection is not anticipated)
* Based on the neurosurgeon's judgment, there is no anticipated physical connection between the post-resection tumor cavity and the cerebral ventricles
* Absolute neutrophil count (ANC) of >= 1500 cells/mm^3
* Platelet count >= 100,000 cells/mm^3
* Total bilirubin =< 2.0 mg/dl
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) =< 4 times the institutional upper limit of normal
* Serum creatinine =< the institutional upper limit of normal
* There is no limit to the number of prior therapies
* Patient must be able to understand and be willing to sign a written informed consent document
* INCLUSION CRITERIA FOR MTD COHORT 2
* Patient has a prior, histopathologically-confirmed diagnosis of glioblastoma
* Patient has not received any therapy for recurrent disease
* INCLUSION CRITERIA FOR PROCEEDING TO TREATMENT WITH IRINOTECAN DURING CYCLE 1
* A patient's daily total dose of dexamethasone must be =< 16 mg by day 3

Exclusion Criteria:

* Patient is homozygous or heterozygous for the UDP glycosyltransferase 1 family, polypeptide A1*28 allele (UGT 1A1*28) allele and/or has Gilbert's disease
* Patient must not be taking any cytochrome P450 3A4 (CYP3A4) hepatic enzyme-inducing anticonvulsants (phenytoin, fosphenytoin [Cerebyx], carbamazepine, phenobarbital, primidone, oxcarbazepine) or other moderate to strong CYP3A4 inhibitors or inducers for at least 2 weeks prior to start of study treatment
* Patient has anti-human leukocyte antigen (HLA) antibodies specific for HLA antigens expressed by the F3.CD.CE NSCs
* Patient has not recovered from any toxicity of prior therapies; an interval of at least 6 weeks must have elapsed since taking a nitrosourea-containing chemotherapy regimen, at least 4 weeks since completing a non-nitrosourea-containing cytotoxic chemotherapy regimen, and at least 2 weeks from taking the last dose of a targeted agent and the start of study treatment, with the exception of bevacizumab, where a wash out period of at least 4 weeks is required before starting study treatment
* Patient is taking flucytosine
* Patient is unable to undergo a magnetic resonance imaging (MRI)
* Patient has chronic or active viral infections of the central nervous system (CNS) or an uncontrolled illness
* Patient may not be receiving any other investigational agents, or concurrent biological, chemotherapy, or radiation therapy
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to irinotecan
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is participating in this study
* A patient with another active malignancy is ineligible for this study
* Non-compliance

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity (DLT), graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | 6 weeks
  Tables will be created to summarize all toxicities and side effects by dose, course, organ severity (by NCI CTCAE version 4.0), and attribution. Rates and associated 95% Clopper Pearson confidence limits will be estimated for the DLT and clinical benefit at the MTD for cohort 1 and cohort 2 and in combination if the results are similar.
Incidence of all attributable toxicities, graded according to NCI CTCAE version 4.0 | Up to 15 years
  Tables will be created to summarize all toxicities and side effects by dose, course, organ severity (by NCI CTCAE version 4.0), and attribution.
Biologic activity of the hCE1m6-NSCs through Cmax and AUC of irinotecan and SN-38 in dialysate and plasma | Prior to the start of the irinotecan infusion and at 90 minutes (just prior to the end of the infusion), and then at 30 minutes, 1, 2, 4, 8, 24, and 48 hours after the end of the infusion on day 3 of week 1
  Data from patients who undergo intracerebral microdialysis will be summarized using descriptive statistics and graphical methods.

SECONDARY OUTCOMES:
Incidence of immunogenicity measured by the development of T cell responses and antibodies against the NSCs using TcR Vβ spectratyping, CD 107 degranulation assays, and flow cytometry | Up to 15 years
  Results will be summarized in an exploratory fashion using descriptive statistics and graphical methods.
NSC biodistribution in the brain via Feraheme-labeling of NSCs and MR imaging | Up to 15 years
  Results will be summarized in an exploratory fashion using descriptive statistics and graphical methods.
Clinical benefit measured by tumor response | Up to 15 years
NSC persistence at autopsy | Up to 15 years
  Results will be summarized in an exploratory fashion using descriptive statistics and graphical methods.

CONTACTS AND LOCATIONS:
Overall Officials: Jana Portnow, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States